CLINICAL TRIAL: NCT03872349
Title: Differential Effects of Saturated and Monounsaturated Fatty Acids on Chylomicron Secretion and Expression of Key Genes That Regulate Intestinal Lipid Metabolism in Insulin Resistant Subjects
Brief Title: Effects of Monounsaturated Fatty Acids on Intestinal Lipid Metabolism in Insulin Resistant Subjects (MUFA )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Patrick Couture, Principal Investigator, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: INAF-MUFA
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monounsaturated fatty acids diet (Experimental): During 4 weeks, subjects eat a diet high in monounsaturated fatty acids (percent of total caloric intake: 15.0% from proteins; 50.0% from carbohydrates; 35.0% from fat: 7.1% from saturated fat; 20.7% from monounsaturated fat; 7.2% from n-6 polyunsaturated fat).
  Interventions: Other: Monounsaturated fatty acids diet; Other: Saturated fatty acids diet
- Saturated fatty acids diet (Experimental): During 4 weeks, subjects eat a diet high in polyunsaturated fatty acids (percent of total caloric intake: 15.0% from proteins; 50.0% from carbohydrates; 35.0% from fat: 13.4% from saturated fat; 14.4% from monounsaturated fat; 7.2% from n-6 polyunsaturated fat).
  Interventions: Other: Monounsaturated fatty acids diet; Other: Saturated fatty acids diet

INTERVENTIONS:
Other: Monounsaturated fatty acids diet — During 4 weeks, subjects eat a diet high in monounsaturated fatty acids and will have a duodenal gastroscopy and a kinetic study at the end of the 4-week period.
Other: Saturated fatty acids diet — During 4 weeks, subjects eat a diet high in saturated fatty acids and will have a duodenal gastroscopy and a kinetic study at the end of the 4-week period.

SUMMARY:
The overaccumulation of apolipoprotein (apo)B-48-containing lipoproteins of intestinal origin observed in patients with insulin-resistance is now thought to be attributable to both elevated intestinal production and reduced clearance of these lipoproteins. Substantial evidence exists indicating that elevated plasma levels of these lipoproteins are associated with increased cardiovascular disease (CVD) risk. Therefore, reduction of atherogenic plasma triglyceride-rich lipoproteins à (TRL) levels of intestinal origin appears to be crucial to improve CVD risk associated with insulin-resistance. In this regard, there is some evidence that the clinical recommendation to replace dietary saturated fatty acids (SFAs) by monounsaturated fatty acids (MUFAs) reduces CVD risk in the general population. Although the beneficial impact of PUFAs on CVD risk has been related primarily to favorable changes in plasma LDL-cholesterol levels, recent data suggest that chronic MUFA consumption may also exert beneficial effects on CVD risk by reducing postprandial lipemia. The impact of substituting SFAs by MUFAs on postprandial lipid response may be of even greater significance in dyslipidemic patients with insulin-resistance among whom intestinal TRLs represent a large proportion of the atherogenic lipoproteins. The general objective of the proposed research is to investigate how dietary MUFAs in place of SFAs modify intestinal lipoprotein metabolism in men and women with dyslipidemia associated with insulin-resistance. The investigators hypothesize that the intestinal secretion of apoB-48-containing lipoproteins will be lower following a diet rich in MUFAs than after consuming a diet rich in SFAs. The investigators also hypothesize that substitution of SFAs by MUFAs will be associated with significant alterations in expression of key genes and proteins involved in intestinal lipoprotein metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18-60 years
* Waist circumference > 102 cm (men) and > 88 cm (women)
* HDL-cholesterol < 1.1 mmol/L (men) and < 1.3 mmol/L (women)
* Triglycerides > 1.7 mmol/L
* Fasting blood glucose > 6.1 mmol/L
* Normal blood pressure (<130/85)

Exclusion Criteria:

* Men and women < 18 or > 60 years
* Smokers (> 1 cigarette/day)
* Body weight variation > 10% during the last 6 months prior to the study baseline
* Subjects with a previous history of cardiovascular disease
* Subjects with type 2 diabetes
* Subjects with a monogenic dyslipidemia
* Subjects on hypertension medications or medications known to affect lipoprotein metabolism or the integrity of gastrointestinal mucosa
* Subjects with endocrine or gastrointestinal disorders
* History of alcohol or drug abuse within the past 2 years
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-09 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Change in TRL apolipoprotein B48 (apoB-48) production rate. | At week 4 and week 12 (at the end of the two 4-weeks diets)

SECONDARY OUTCOMES:
Changes in duodenal expression of Niemann-Pick C1-like 1, Adenosine triphosphate-binding cassette transporters, Fatty Acid Binding Protein, Sterol Regulatory Element Binding Protein. | At week 4 and week 12 (at the end of the two 4-weeks diets)
Changes in duodenal expression of diacylglycerol acyltransferase, Acyl-CoA:cholesterol O-acyltransferase 2 and 3-hydroxy-methylglutaryl-CoA reductase. | At week 4 and week 12 (at the end of the two 4-weeks diets)
Change in synthesis of apoB-48 containing lipoproteins (Microsomal triglyceride transfer protein (MTP), apoB-48). | At week 4 and week 12 (at the end of the two 4-weeks diets)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, FRCP, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desjardins LC, Briere F, Tremblay AJ, Rancourt-Bouchard M, Drouin-Chartier JP, Corbeil J, Lemelin V, Charest A, Schaefer EJ, Lamarche B, Couture P. Substitution of dietary monounsaturated fatty acids from olive oil for saturated fatty acids from lard increases low-density lipoprotein apolipoprotein B-100 fractional catabolic rate in subjects with dyslipidemia associated with insulin resistance: a randomized controlled trial. Am J Clin Nutr. 2024 May;119(5):1270-1279. doi: 10.1016/j.ajcnut.2024.03.015. Epub 2024 Mar 20. PMID 38518848